CLINICAL TRIAL: NCT07331038
Title: Longitudinal Assessment of Postoperative Muscle Loss and Nutritional Status After Gastrectomy
Brief Title: Postoperative Muscle Loss After Gastrectomy
Status: Not yet recruiting | Type: Observational
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 202511030RIND
Record Dates: First submitted 2025-12-28; First posted 2026-01-09 (Actual); Last update posted 2026-01-09 (Actual); Status verified 2025-12

CONDITIONS: Postoperative Muscle Loss
Keywords: postoperative muscle loss

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Biospecimen Retention: Samples With DNA — for investigating nutrition gene condition
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Investigating postoperative muscle loss after gastrectomy

DETAILED DESCRIPTION:
Surgical-related muscle loss (SRML) is a common postoperative complication, defined as a reduction of at least 10% in preoperative skeletal muscle mass in at least one upper limb and one lower limb by postoperative day 7. Patients undergoing gastric cancer surgery are typically older and at high risk for low muscle mass, and surgical stress further exacerbates the incidence of SRML. In addition to limb skeletal muscles, swallowing-related muscle groups may also be affected, leading to impaired nutritional intake and increased risks of postoperative complications and mortality. In recent years, ultrasonography-owing to its noninvasiveness, bedside feasibility, and repeatability-has been regarded as a practical tool for monitoring postoperative muscle changes. This study aims to longitudinally track changes in skeletal muscle thickness using ultrasound in patients undergoing gastrectomy for gastric cancer, while concurrently assessing nutritional status and clinical recovery, with the goal of establishing an early clinical assessment model for detecting postoperative muscle loss to inform nutritional interventions and postoperative care. Accordingly, this project will conduct a cohort study of 100 patients to investigate postoperative muscle loss and associated risk factors, including swallowing function and postoperative complications. This prospective observational study will enroll patients aged ≥20 years who undergo gastrectomy and provide written informed consent; individuals with psychiatric conditions that may impair consent or study procedures will be excluded. A total of 100 patients undergoing gastric cancer resection will be assessed preoperatively (T0) and at postoperative day 7 ±2 (T1), 1 month ±1 week (T2), 3 months ±2 weeks (T3), 6 months ±2 weeks (T4), and 12 months ±2 weeks (T5). Assessments will include ultrasound-measured muscle thickness, bioelectrical impedance analysis, handgrip strength and limb muscle strength, tongue pressure, life quality and activity associated questionnaire, and blood tests for nutritional, markers. The expected outcome is that patients with lower preoperative muscle mass and those at high risk of malnutrition will be more susceptible to postoperative muscle loss, and the occurrence of postoperative muscle loss will be associated with an increased risk of postoperative complications.

ELIGIBILITY:
Inclusion Criteria:

* gastrectomy

Exclusion Criteria:

* unable to follow our order

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patients undergoing gastrectomy
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2025-12-12 (Estimated); Primary Completion 2030-12-31 (Estimated); Study Completion 2031-12-31 (Estimated)

PRIMARY OUTCOMES:
surgical related muscle loss | follow up to postoperative 1 year
  four limb muscle thickness measurement